CLINICAL TRIAL: NCT03374215
Title: Clinical and Molecular Characteristics of Primary Aldosteronism in Blacks
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180031; 18-CH-0031
Record Dates: First submitted 2017-12-14; First posted 2017-12-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-07-17

CONDITIONS: Adrenal Gland Neoplasm; Hypertension; Bone Diseases, Metabolic; Cardiovascular Disease; Hyperinsulinemia
Keywords: Adrenal Adenoma; Molecular Genetics; African-American; Biomarkers; Primary Aldosteronism; Natural History
MeSH Terms: conditions — Adrenal Gland Neoplasms; Hypertension; Bone Diseases, Metabolic; Cardiovascular Diseases; Hyperinsulinism; ACTH Syndrome, Ectopic; Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult AA with primary aldosteronism: Adult individuals (age 18 or older) with HTN and discrete adrenal masses or bilateral hyperplasia of the adrenal glands, with outpatient positive ARR or string clinical suspicion for PA
- Family members age >= 7 of participants: DNA from relatives of patients (age 7 or older)

SUMMARY:
Background:

The adrenal gland makes the hormone aldosterone. This helps regulate blood pressure. An adrenal gland tumor that makes too much aldosterone can cause high blood pressure and low potassium. The cause of these tumors is unknown, but sometimes they are inherited.

Objective:

To study the genes that may cause primary aldosteronism in Black individuals.

Eligibility:

People ages 18-70 who:

Are Black, African American, or of Caribbean descent

And have difficult to control blood pressure or primary aldosteronism

Relatives of people with primary aldosteronism

Design:

Participants who are relatives of people with primary aldosteronism will have only 1 visit, with medical history and blood tests.

Participants with primary aldosteronism or difficult to control blood pressure (suspected to possibly have primary aldosteronism) will be screened with a 1-2 hour visit. If they qualify, they will return for a hospital stay for 7-10 days. Tests may include:

Medical history

Physical exam

Blood tests: Participants will have a small tube (IV catheter) inserted in a vein in the arm. They may drink a glucose-containing liquid or get a salt solution. If medically indicated, they may have invasive blood tests with a separate consent.

Urine tests: Some require a high-salt diet for 3 days.

Heart tests

Scans: Participants lie in a machine that takes pictures of the body. A dye may be injected through a vein.

Small hair sample taken from near the scalp.

Kidney ultrasound

Bone density scan: Participants lie on a table while a camera passes over the body.

If the doctors feel it is medically necessary, they will offer participants treatment depending on their results. These treatments may cure the patient of their disease and may include:

1. Having one adrenal gland removed by the Endocrine surgeon under anesthesia. Patients will have follow-up visits 2-4 weeks after surgery.
2. Taking drugs to block the effects of aldosterone

Participants may return about 1 year later to repeat testing.

DETAILED DESCRIPTION:
Primary Aldosteronism (PA) is the most common cause of secondary hypertension, accounting for 6-8% of hypertension and 14-25% of resistant hypertension. This prevalence translates to approximately 1 in 30-50 adults or about 4,000,000 Americans with PA. Until recently, the deleterious effects of PA were thought to derive solely from aldosterone-mediated sodium retention and associated blood pressure rise. However, animal studies and clinical trials demonstrate that mineralocorticoid receptor (MR) blockade has cardio- and reno-protective effects that clearly exceed those expected from blood pressure reduction alone. Growing evidence supports the concept that excess aldosterone, in the presence of elevated blood pressure, initiates a cascade characterized by fibrosis, oxidative stress, and activation of pro-inflammatory and pro-fibrotic pathways, leading to morbidity via worsened insulin sensitivity, impaired bone formation, and accelerated cardiovascular remodeling. Recent studies have identified several new genetic underpinnings of PA, both germline and somatic, including mutations in KCNJ5, ATP1A1, ATP2B3, CACNA1D, and ARMC5. As the effects of chronic hyperaldosteronism differ between races, it is not surprising that the relative prevalence of these mutations differs among cohorts. African Americans (AA) in particular have increased susceptibility to end-organ damage from aldosterone excess-induced cardiovascular remodeling. They are more likely to have congestive heart failure, end-stage renal disease, and atherosclerotic events than age-matched Caucasians. However, to date no comprehensive analysis of mutations in PA has been performed in AA. (Note: for the purposes of this protocol, the terms Black or African American incorporate individuals who self-identify as Black, African American, or the Caribbean diaspora).

The aims of this study are to identify the germline and/or somatic mutations causing PA in AA, define the effects of these mutations on aldosterone production in AA, and to identify effective pharmacologic agents that will inhibit inappropriate aldosterone production in target cells. Aldosterone producing adenoma (APA) and other adrenocortical tumor (ACT) specimens will be gathered from archival (collected under protocol 00-CH-160 and other related NIH studies) and prospective research subjects with PA that will be evaluated at the NIH Clinical Research Center under the proposed protocol. Samples will be analyzed using state-of-the-art next-generation sequencing (NGS). Human adrenal cell lines (H295R and others, as appropriate) will be used to study the mutations effect on aldosterone production. Additionally, this will help identify possible effective pharmacologic therapeutics to treat PA. Animal models of novel genetic causes of PA may also be created to study the molecular mechanisms underpinning the disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for main study:

* Age greater than or equal to 18y.
* Self-described Black race. Those with reported other racial backgrounds may enroll in protocol 00-CH-0160 instead.
* Evidence supportive of the diagnosis of PA (e.g. HTN, hypokalemia, known adrenal nodule, elevated ARR, etc).
* Willing and able to return to the NIH for follow-up evaluation.

Inclusion criteria for blood (peripheral) DNA only study:

* Age greater than or equal to 7y.
* Relative of a patient that participates in the main study (above) (i) with family history of hypertension, ACTs, or both, or (ii) with a genetic mutation identified in the course of the genetic investigations described in the main study.

EXCLUSION CRITERIA:

Exclusion criteria for main study:

* Individuals over the age of 70 years will be excluded because of the possibility of comorbidities that may significantly affect appropriate initial work-up and post-operative management. In addition, research data may be compromised by the inability to interpret data collected from patients over the age of 70 years that may be on multiple medications for a variety for reasons.
* Women who are pregnant or nursing will be excluded for safety concerns with hyperaldosteronism workup.
* Individuals whose medical status will not allow them, for safety reasons, to participate in the provocative testing (e.g. NYHA Class III or IV heart failure, or CKD Stage 3b or worse), or who in the opinion of the investigators have unacceptably high risk for surgical morbidity and mortality (e.g. Revised Cardiac Risk Index Class IV or above, or American Society of Anesthesiologists Physical Status Class 3 or above) will be excluded from the protocol, as they will not be able to participate profitably in the research aspects of this protocol.
* Individuals who have current substance abuse or a psychiatric disorder or any other condition that in the opinion of the investigators would impede competence, compliance, or participation in the study.
* Individuals found to have a known inherited syndrome as the cause for hormone over-secretion will be excluded from participation in this protocol, as the mechanisms of hormone over-secretion and tumorigenesis is likely to be distinct in these individuals. Specific examples of syndromes that may be excluded from this protocol include individuals with Carney complex, McCune-Albright syndrome, and MEN-1. If inquiries are received from such patients, they will be referred to the appropriate ongoing protocols, if possible.
* Family members who end up being diagnosed with PA will be referred to the 00-CH-0160 protocol, to avoid selection bias in genetic mutation analyses for PA.
* Patients unwilling or unable to abide by procedures of the protocol.

<TAB>

Exclusion criteria for the DNA only study:

-Patients unwilling or unable to provide peripheral blood for DNA studies.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical, referrals from community physicians@@@
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To define the germline and/or somatic genetic events causing Primary Aldosteronism (PA) in Blacks. | baseline, end of study
  define the causes of PA in AA and develop new therapeutic strategies to inhibit the inappropriate aldosterone production.
To define the effects of mutations in Black subjects on adrenocortical tumor formation, function and aldosterone production. | Continuous
  define the causes of PA in AA and develop new therapeutic strategies to inhibit the inappropriate aldosterone production.

SECONDARY OUTCOMES:
To investigate the clinical utility of other biomarkers in the subtype classification of PA. | baseline, end of study
  define the causes of PA in AA and develop new therapeutic strategies to inhibit the inappropriate aldosterone production.
To investigate the cardiovascular, renal, metabolic, bone, and coagulopathic consequences of PA in AA, as well as any changes after one year of directed therapeutic intervention (e.g. post-adrenalectomy or mineralocorticoid receptor antagonist t... | baseline, end of study
  define the causes of PA in AA and develop new therapeutic strategies to inhibit the inappropriate aldosterone production.
To investigate co-secretion of other steroids in PA. | baseline, end of study
  define the causes of PA in AA and develop new therapeutic strategies to inhibit the inappropriate aldosterone production.

CONTACTS AND LOCATIONS:
Overall Officials: Sanaz Sakiani, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-CH-0031.html